CLINICAL TRIAL: NCT00286273
Title: Safety and Efficacy of the Use of Regional Anticoagulation With Citrate in Continuous Venovenous Hemofiltration, a Randomized Controlled Trial Comparing Anticoagulation With Citrate to the Low Molecular Weight Heparin Nadroparin
Brief Title: Safety and Efficacy of the Use of Regional Anticoagulation With Citrate in Continuous Venovenous Hemofiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: HM Oudemans-van Straaten, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WON 03.1
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Kidney Failure, Acute
Keywords: kidney failure, acute; venovenous hemofiltration; hemorrhage; heparin, low-molecular-weight; nadroparin; citrates
MeSH Terms: conditions — Acute Kidney Injury; Hemorrhage | interventions — trisodium citrate; Citric Acid; Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- citrate (Active Comparator): regional anticoagulation with citrate
  Interventions: Drug: trisodium citrate
- nadroparin (Active Comparator): nadroparin is a low molecular weight heparin
  Interventions: Drug: nadroparin

INTERVENTIONS:
Drug: trisodium citrate — for regional anticoagulation of the extracorporeal CVVH circuit
  Other Names: regional anticoagulation with citrate
  Arms: citrate
Drug: nadroparin — for anticoagulation of the extracorporeal CVVH circuit
  Other Names: nadroparin is a low molecular weight heparin
  Arms: nadroparin

SUMMARY:
Severely ill patients admitted to the intensive care unit may develop an acute failure of kidney function. To bridge the period to recovery, renal function is temporarily replaced by continuous venovenous hemofiltration (CVVH). To prevent clotting of the hemofiltration circuit, heparin is generally used, providing anticoagulation in the circuit and the patient. As a result, bleeding complications may occur, necessitating the transfusion of blood. Anticoagulation of the circuit can also be obtained with the use of tri-sodium citrate, which provides anticoagulation of the circuit without affecting coagulation in the patient and thus without increasing his/her risk of bleeding. The use of citrate may however cause metabolic complications.

Primary aim of the present study is to show in a larger group of intensive care patients whether the use of regional anticoagulation with citrate is safe compared to systemic anticoagulation with the low molecular weight heparin nadroparin.

DETAILED DESCRIPTION:
Severely ill patients admitted to the intensive care unit may develop an acute failure of kidney function. Renal function generally recovers if the acute illness improves. To bridge this period, renal function is temporarily replaced by continuous hemofiltration, so called continuous venovenous hemofiltration (CVVH). To remove toxic substances and fluids, the patient's blood flows through a circuit, containing a filter. Flow in the filter is regulated by the CVVH-device.

Normally blood starts to clot as soon as it leaves the body. To prevent clotting of the blood in the filter, the blood has to be 'anticoagulated'. For this purpose, heparins are generally used. Heparins make the blood less likely to clot. Drawback of the use of heparins is that they not only prevent clotting of blood in the circuit and the filter, but also in the patient. Heparins thereby increase the risk of bleeding. Intensive care patients are at higher risk of bleeding due to a recent operation or trauma, ulcers in the mouth or the stomach, or abnormalities in their blood to the acute illness. Due to the continuous application of CVVH for days, anticoagulation is administered without interruption over prolonged periods of time. Studies report bleeding complications in 5 to 50% of the patients. As a result of bleeding, patients need blood transfusion and sometimes surgery. Control of bleeding is sometimes extremely difficult.

An alternative to heparin is citrate, which allows regional anticoagulation of the circuit and the filter without an effect increasing the risk of bleeding for the patient. Anticoagulation with citrate is more complex, nurses need to follow a strict protocol.. Several small studies have shown that regional anticoagulation with citrate is associated with less bleeding and a longer filter survival. The use if citrate is however associated with a greater risk of metabolic complications, if the protocol is not strictly followed. Primary aim of the present study is to show in a larger group of intensive care patients whether the use of regional anticoagulation with citrate is safe compared to systemic anticoagulation with the low molecular weight heparin nadroparin.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care patients scheduled for continuous venovenous hemofiltration

Exclusion Criteria:

* Severe pre-existent liver failure (cirrhosis Child C), acute liver dysfunction as occurring with septic shock is not a reason for exclusion
* Active bleeding or bleeding necessitating the infusion of two red blood cell units within 24 hours before starting hemofiltration or a fall in hemoglobin of > 0.5 mmol/l. A fall in hemoglobin/hematocrit as a result of fluid loading is not regarded as bleeding.
* Surgery within 24 h prior to CVVH.
* Patients needing full systemic anticoagulation (unfractionated heparin in a dose of > 10000 IU/day, or nadroparin > 3800 IU/day) for other reasons
* Expectation to die within 24 hours
* Chronic dialysis
* Proven or suspected heparin-induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2003-03; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
bleeding complications | during administration of study anticoagulant
transfusion requirement | during administration of study anticoagulant
filter survival | during hemofiltration

SECONDARY OUTCOMES:
mortality | 3-month and hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Heleen M Oudemans-van Straaten, MD,PhD, Principal Investigator — Onze Lieve Vrouwe Gasthuis
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands

REFERENCES:
- [Result] Oudemans-van Straaten HM, Bosman RJ, Koopmans M, van der Voort PH, Wester JP, van der Spoel JI, Dijksman LM, Zandstra DF. Citrate anticoagulation for continuous venovenous hemofiltration. Crit Care Med. 2009 Feb;37(2):545-52. doi: 10.1097/CCM.0b013e3181953c5e. PMID 19114912
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078